CLINICAL TRIAL: NCT01858571
Title: Low Dose Chemotherapy (Metronomic Therapy) Versus Best Supportive Care in Progressive and/or Refractory Pediatric Malignancies: a Double Blind Placebo Controlled Randomized Study
Brief Title: Low Dose Chemotherapy Versus Best Supportive Care in Progressive Pediatric Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sameer Bakhshi, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEC/NP-63/2013
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Malignant Childhood Neoplasm
Keywords: Childhood Cancer
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose chemotherapy (Experimental): Alternating cycles of Cycle A and B (Each cycle includes 3 weeks of drug administration) with each drug rounded off to the nearest tablet/capsule size.
  Cycle A
  * Daily oral Thalidomide (at 3mg/kg)
  * Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
  * Daily oral Etoposide (50 mg/m2/d)
  Cycle B
  * Daily oral Thalidomide (at 3mg/kg)
  * Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
  * Daily oral Cyclophosphamide (2.5 mg/kg/d to a maximum of 100 mg/d) every 21 days
  Interventions: Drug: Low dose chemotherapy
- Best supportive care (Placebo Comparator): Placebo: Alternating cycles of Cycle A and B (Each cycle includes 3 weeks of drug administration)
  * Capsules of same size and color as used in metronomic therapy Best supportive care
  * Management of pain as per WHO standard for pain management
  Interventions: Drug: Low dose chemotherapy

INTERVENTIONS:
Drug: Low dose chemotherapy — Metronomic chemotherapy schedule : Alternating cycles of Cycle A and B (Each cycle includes 3 weeks of drug administration) with each drug rounded off to the nearest tablet/capsule size.
  Cycle A
  * Daily oral Thalidomide (at 3mg/kg)
  * Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
  * Daily oral Etoposide (50 mg/m2/d)
  Cycle B
  * Daily oral Thalidomide (at 3mg/kg)
  * Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
  * Daily oral Cyclophosphamide (2.5 mg/kg/d to a maximum of 100 mg/d) every 21 days
  Other Names: •Thalidomide •Celecoxib •Etoposide •Cyclophosphamide

SUMMARY:
Many of the pediatric malignancies are not curable on progression on front line or 2nd line chemotherapy. Further therapy with conventional drugs imposes many side effects and decreases the QOL. The usual therapy offered to such patients is best supportive care.

Metronomic chemotherapy can induce tumor stabilization or tumor responses in patients with cancer that are refractory or have relapsed after conventional chemotherapy. Whether metronomic therapy is better than best supportive care is not known. In order to do so, a study is required which may compare metronomic therapy with a placebo therapy on PFS and QOL in relapsed refractory cases of pediatric solid tumors who have failed at least two lines of chemotherapy.

HYPOTHESIS

The investigators hypothesize that metronomic chemotherapy in progressive pediatric malignancy will improve PFS and QOL. If validated, then this form for therapy will be an option for both the patients and the clinicians, who are left with just an option of best supportive care in such situations of progressive pediatric cancers despite multiple lines of chemotherapy.

DETAILED DESCRIPTION:
Many of the pediatric malignancies are not curable on progression on front line or 2nd line chemotherapy. Further therapy with conventional drugs imposes many side effects and decreases the QOL. The usual therapy offered to such patients is best supportive care.

Metronomic chemotherapy can induce tumor stabilization or tumor responses in patients with cancer that are refractory or have relapsed after conventional chemotherapy. Whether metronomic therapy is better than best supportive care is not known. In order to do so, a study is required which may compare metronomic therapy with a placebo therapy on PFS and QOL in relapsed refractory cases of pediatric solid tumors who have failed at least two lines of chemotherapy.

It will be double blind randomized study. One group will receive metronomic therapy along with best supportive care and other will receive placebo and best supportive care.

The treatment will be continued till progression is documented. Metronomic chemotherapy schedule : Alternating cycles of Cycle A and B (Each cycle includes 3 weeks of drug administration) with each drug rounded off to the nearest tablet/capsule size.

Cycle A

* Daily oral Thalidomide (at 3mg/kg)
* Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
* Daily oral Etoposide (50 mg/m2/d) Cycle B
* Daily oral Thalidomide (at 3mg/kg)
* Daily oral Celecoxib (100 mg BID for patients < 20 kg, 200 mg BID for patients 20-50 kg, and 400 mg BID for patients > 50 kg)
* Daily oral Cyclophosphamide (2.5 mg/kg/d to a maximum of 100 mg/d) every 21 days

Placebo: Alternating cycles of Cycle A and B (Each cycle includes 3 weeks of drug administration)

* Capsules of same size and color as used in metronomic therapy Best supportive care
* Management of pain as per WHO standard for pain management

The dose of medications in capsules have to be rounded off to the nearest capsule size. Instead of rounding off on the daily dose, the total dose over the week would be calculated and rounded off and divided over 5-6 days in a week. This is being done so as to prevent any extra dosing.

If any grade 3-4 toxicity occurs in the first course, then the dose for chemotherapy would be reduced in the subsequent course by 20%.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory/Progressive non hematopoietic extracranial solid tumors following treatment with at least 2 lines of chemotherapy.
2. ECOG performance status (<=3)(at least patients ambulating with crutches or on wheel chair)
3. Age: 5-18 years
4. Recovered from all acute toxic effects of earlier therapy
5. Absolute neutrophil count > 1X 109/L
6. Absolute platelet count > 75 x 109/L
7. Normal renal functions
8. Serum bilirubin <1.5 times the upper limit of normal, and the serum aspartate aminotransferase and alanine aminotransferase < 5 times the upper limit of normal.

Exclusion Criteria:

1. Uncontrolled concurrent illness or active infection
2. Positive serology for human immunodeficiency.
3. Unable to swallow oral medication
4. Pregnant and breast-feeding

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to 2 years

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years

OTHER OUTCOMES:
Quality of life | Up to 2 years
Bio marker of angiogenesis (VEGF) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Bakhshi, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Pramanik R, Agarwala S, Sreenivas V, Dhawan D, Bakhshi S. Quality of life in paediatric solid tumours: a randomised study of metronomic chemotherapy versus placebo. BMJ Support Palliat Care. 2023 Jun;13(2):234-237. doi: 10.1136/bmjspcare-2020-002731. Epub 2021 Jan 19. PMID 33468507
- [Derived] Pramanik R, Agarwala S, Gupta YK, Thulkar S, Vishnubhatla S, Batra A, Dhawan D, Bakhshi S. Metronomic Chemotherapy vs Best Supportive Care in Progressive Pediatric Solid Malignant Tumors: A Randomized Clinical Trial. JAMA Oncol. 2017 Sep 1;3(9):1222-1227. doi: 10.1001/jamaoncol.2017.0324. PMID 28384657